CLINICAL TRIAL: NCT00002701
Title: INDUCTION WITH ALL-TRANS RETINOIC ACID IN COMBINATION WITH IDARUBICIN AND INTENSIVE CONSOLIDATION FOLLOWED BY BONE MARROW TRANSPLANTATION OR A RANDOMIZED MAINTENANCE TREATMENT DEPENDING UPON THE AMOUNT OF MINIMAL RESIDUAL DISEASE IN ACUTE PROMYELOCYTIC LEUKEMIA
Brief Title: Combination Chemotherapy With or Without Bone Marrow Transplantation in Treating Patients With Acute Promyelocytic Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064499; EORTC-06952; ITA-GIMEMA-AIEOP-1
Record Dates: First submitted 1999-11-01; First posted 2003-04-11 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2006-11

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; adult acute promyelocytic leukemia (M3)
MeSH Terms: conditions — Leukemia; Leukemia, Promyelocytic, Acute | interventions — Busulfan; Cyclophosphamide; Cytarabine; Etoposide; Idarubicin; Mercaptopurine; Methotrexate; Mitoxantrone; Thioguanine; Tretinoin; Radiotherapy

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Drug: cytarabine
Drug: etoposide
Drug: idarubicin
Drug: mercaptopurine
Drug: methotrexate
Drug: mitoxantrone hydrochloride
Drug: thioguanine
Drug: tretinoin
Procedure: allogeneic bone marrow transplantation
Procedure: autologous bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy to kill tumor cells. It is not yet known which regimen of combination chemotherapy with or without bone marrow transplantation is more effective in treating promyelocytic leukemia

PURPOSE: Randomized phase III trial to compare the effectiveness of different combination chemotherapy regimens with or without bone marrow transplantation in treating patients who have promyelocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete remission (CR) rate in patients with acute promyelocytic leukemia treated with induction comprising tretinoin (ATRA) and idarubicin (IDA).
* Determine the presence of the promyelocyte-retinoic acid receptor alpha (PML-RARa) transcript using polymerase chain reaction (PCR) in patients with CR after 3 sequential consolidation regimens comprising cytarabine (ARA-C) plus IDA, followed by mitoxantrone plus etoposide, and then IDA, ARA-C, and thioguanine.
* Determine the percentage of patients who complete the protocol, including PML-RARa-positive patients treated with post-consolidation bone marrow transplantation (BMT) and PML-RARa-negative patients treated with maintenance comprising mercaptopurine (MP) plus methotrexate (MTX) vs ATRA only vs MP plus MTX alternating with ATRA vs observation only.
* Compare the disease-free survival (DFS) and overall survival of these patients treated with these regimens.
* Determine the rate and type of grade 4 toxicity, treatment-related mortality, and time to granulocyte and platelet recovery associated with each phase of treatment in these patients.
* Determine the DFS and overall survival of PML-RARa-positive patients who are ineligible for BMT and are treated with maintenance comprising MP plus MTX alternating with ATRA.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study.

* Induction: Patients receive oral tretinoin (ATRA) twice daily beginning on day 1 and continuing for 30-90 days and idarubicin (IDA) IV over 15 minutes on days 2, 4, and 8. ATRA is discontinued before day 90 in the presence of complete remission (CR) at day 30 or 60, unacceptable toxicity, or disease progression or in the absence of at least a partial remission at day 60. Patients who achieve CR during induction proceed to consolidation.
* Consolidation:

  * First consolidation: Within 2 weeks after achieving CR, patients receive cytarabine (ARA-C) IV over 6 hours followed 3 hours later by IDA IV over 15 minutes on days 1-4.
  * Second consolidation:Within 4-6 weeks after initiation of first consolidation, patients receive mitoxantrone IV over 30 minutes and etoposide IV over 1 hour (beginning 12 hours after initiation of mitoxantrone infusion) on days 1-5.
  * Third consolidation:Within 4-6 weeks after initiation of second consolidation, patients receive ARA-C subcutaneously every 8 hours and oral thioguanine every 8 hours on days 1-5 and IDA IV over 15 minutes on day 1.

Patients proceed to group A if they are promyelocyte-retinoic acid receptor alpha (PML-RARa)-negative after recovery from third consolidation. Patients proceed to allogeneic bone marrow transplantation (BMT) on group B if they are PML-RARa-positive, achieve CR, are under age 55, and have an HLA-A, -B, and -DR identical, chronic myelomonocytic leukemia nonreactive, family donor after recovery from third consolidation. Patients proceed to autologous BMT on group B if they are PML-RARa-positive, achieve CR, and have no identical family donor or are age 55 and over after recovery from third consolidation. Patients proceed to arm III of group A if they are PML-RARa-positive and ineligible for BMT after recovery from third consolidation.

* Group A (maintenance): Patients are stratified according to participating center and initial white blood cell count. Patients are randomized to 1 of 4 treatment arms.

  * Arm I: Patients receive oral mercaptopurine (MP) daily and oral methotrexate (MTX) weekly.
  * Arm II: Beginning 3 months after recovery from third consolidation, patients receive oral ATRA on days 1-15.

Treatment on arms I and II continues every 3 months for 2 years in the absence of disease progression or unacceptable toxicity.

* Arm III: Patients receive 1 course of arm I treatment, alternated by 1 course of arm II treatment. Alternating treatment continues every 3 months for 2 years in the absence of disease progression or unacceptable toxicity.
* Arm IV: Patients undergo observation only.

  * Group B: Eligible patients receive conditioning comprising cyclophosphamide (CTX) IV for 2 days followed by total body irradiation or oral busulfan on days -9 to -6 and CTX on days -5 to -2. Autologous or allogeneic bone marrow is infused on day 0 (within 4 months after initiation of third consolidation).

Quality of life is assessed at baseline, after induction, after each consolidation regimen, and then every 3 months beginning after treatment on group A or B.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 750 patients will be accrued for this study within 7.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute promyelocytic leukemia
* Must have promyelocyte-retinoic acid receptor alpha transcript at disease presentation

PATIENT CHARACTERISTICS:

Age:

* 16 to 74

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 3 times upper limit of normal (ULN)
* AST no greater than 3 times ULN
* Alkaline phosphatase no greater than 3 times ULN

Renal:

* Creatinine no greater than 2.5 mg/dL

Cardiovascular:

* No cardiac contraindication to anthracycline chemotherapy

Other:

* No active serious infection not controlled by antibiotics
* No severe concurrent psychiatric disease
* No other malignancy except basal cell carcinoma
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No concurrent cytotoxic chemotherapy

Endocrine therapy:

* Prior corticosteroids for leukemia allowed

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No prior antileukemic therapy

Ages: 16 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 1995-10

CONTACTS AND LOCATIONS:
Overall Officials: Petra Muus, MD, PhD, Study Chair — Universitair Medisch Centrum St. Radboud - Nijmegen; Franco Mandelli, MD, Study Chair — Azienda Policlinico Umberto Primo
Locations (71):
- Innsbruck Universitaetsklinik, Innsbruck, Austria
- Belgium (9):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - A.Z. St. Jan, Bruges
  - Hopital Universitaire Erasme, Brussels
  - C.H.U. Saint-Pierre, Brussels (Bruxelles)
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
  - CHU Sart-Tilman, Liège
  - Centre Hospitalier Peltzer-La Tourelle, Verviers
- Croatia (2):
  - University Hospital Rebro, Zagreb
  - Medical School/University of Zagreb, Zagreb (Agram)
- Onkologicka Klinka A Onkologicka Lab, Prague, Czechia
- France (7):
  - Centre Hospitalier Regional de Lille, Lille
  - Hopital Edouard Herriot, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hotel Dieu de Paris, Paris
  - Hopital Necker, Paris
  - Centre Medico-Chirurgical Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Klinikum Duisburg, Duisburg
  - Klinikum Grosshadern, Munich (Muenchen)
- Italy (41):
  - Ospedale Civile Alessandria, Alessandria
  - Ospedale Torrette University Ancona, Ancona
  - Ospedale Civile Avellino, Avellino
  - Universita Degli Studi di Bari Policlinico, Bari
  - Ospedale Regionale A. Di Summa, Brindisi
  - Ospedale Oncologico A. Businco, Cagliari
  - Ospedale Ferrarotto, Catania
  - Ospedale Regionale A. Pugliese, Catanzaro
  - Centro Trapianti di Midollo Osseo, Cremona
  - Ospedale Santa Croce, Cuneo
  - Policlinico di Careggi, Firenze (Florence)
  - Ospedali Riuniti Foggia, Foggia
  - Ospedale S. Antonio Abate, Gallarate Varese
  - Ospedale San Martino/Cliniche Universitarie Convenzionate, Genoa (Genova)
  - Ospedale Gen. Provinciale Santa Maria Goretti, Latina
  - Ospedale Maggiore Lodi, Lodi
  - Istituto Scientifico H.S. Raffaele, Milan
  - Ospedale Maggiore Ca Granda, Milano (Milan)
  - Ospedale Di Montefiascone, Montefiascone
  - Azienda Ospedaliera "A. Cardarelli", Naples (Napoli)
  - Federico II University Medical School, Naples (Napoli)
  - Ospedale S. Gennora USL 42, Naples (Napoli)
  - Ospedale Nuovo Pellegrini, Naples (Napoli)
  - Ospedale San Francesco, Nuoro
  - Azienda Ospedaliera di Padova, Padova (Padua)
  - Policlinico - Cattedra di Ematologia, Palermo
  - Ospedale Cervello, Palermo
  - Azienda Ospedaliera Di Parma, Parma
  - I.R.C.C.S. Policlinico San Matteo, Pavia
  - Policlinico Monteluce, Perugia
  - Ospedale San Salvatore, Pesaro
  - Ospedale Civile Pescara, Pescara
  - Ospedale San Carlo, Potenza
  - Ospedale San Eugenio, Rome
  - Azienda Policlinico Umberto Primo, Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Istituto di Ematologia Universita - University di Sassari, Sassari
  - Ospedal SS Annunziata, Taranto
  - Cattedra di Immunologia Clinica, Turin (TO)
  - Ospedale Molinette, Turin (Torino)
- Netherlands (7):
  - Leyenburg Ziekenhuis, 's-Gravenhage (Den Haag, the Hague)
  - Groot Ziekengasthuis 's-Hertogenbosch, 's-Hertogenbosch
  - Academisch Medisch Centrum, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen
  - University Hospital - Rotterdam Dijkzigt, Rotterdam
- Ibn-i Sina Hospital, Ankara University, Ankara, Turkey (Türkiye)